CLINICAL TRIAL: NCT07279558
Title: Effects of Full-spectrum Cannabidiol on Alcohol Consumption and Alcohol Use Disorder Phenotypes: Implications for Precision Medicine
Brief Title: Cannabidiol and Alcohol Use Disorder Phenotypes
Acronym: CAP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-1612; R01AA031664 (NIH)
Record Dates: First submitted 2025-12-10; First posted 2025-12-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Cannabidiol
MeSH Terms: conditions — Alcoholism | interventions — hempseed oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Full-Spectrum CBD (Experimental): Subjects will take 200 mg of full-spectrum CBD ([fsCBD] CBD that contains <0.3% THC) daily for 8 weeks. The total dose is split into a morning and evening dose, such that participants in the fsCBD condition will take approximately 100mg fsCBD in the morning (2 capsules) and 100mg fsCBD in the evening (2 capsules).
  Interventions: Drug: Full-Spectrum Cannabidiol (CBD)
- Broad- Spectrum CBD (Experimental): Subjects will take 200 mg of broad-spectrum CBD ([bsCBD] CBD that contains no THC) daily for 8 weeks. The total dose is split into a morning and evening dose, such that participants in the bsCBD condition will take approximately 100mg bsCBD in the morning (2 capsules) and 100mg bsCBD in the evening (2 capsules).
  Interventions: Drug: Broad-Spectrum Cannabidiol (CBD)
- Placebo (Placebo Comparator): Subjects will take a matching placebo solution (100% Hemp Seed Oil) daily for 8 weeks. The total dose is split into a morning and evening dose, such that participants in the condition will take approximately 100mg hemp seed oil in the morning (2 capsules) and 100mg hemp seed oil in the evening (2 capsules).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Full-Spectrum Cannabidiol (CBD) — Dose: Approximately 200mg of full-spectrum CBD (<0.3% THC) Active Ingredients: Full spectrum hemp extract Other Ingredients: Hemp seed oil, glycerin, gelatine.
  Other Names: Hemp-derived, full-spectrum cannabidiol; Ecofibre USA/Ananda Hemp
  Arms: Full-Spectrum CBD
Drug: Broad-Spectrum Cannabidiol (CBD) — Dose: Approximately 200mg of broad-spectrum CBD, (0% THC) Active Ingredients: Broad spectrum hemp extract Other Ingredients: Hemp seed oil, glycerin, gelatine.
  Other Names: Hemp-derived, broad-spectrum cannabidiol; Ecofibre USA/Ananda Hemp
  Arms: Broad- Spectrum CBD
Drug: Placebo — Active Ingredients: N/A Other Ingredients: Hemp seed oil, glycerin, gelatine.
  Other Names: 100% Hemp Seed Oil; Ecofibre USA/Ananda Hemp
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare the effects of Full-Spectrum CBD (CBD containing a small amount of THC), Broad-Spectrum CBD (CBD with no THC), and placebo on alcohol consumption and clinically relevant Alcohol Use Disorder (AUD) phenotypes among adults with AUD. The main questions it aims to answer are:

* Does Full-Spectrum CBD (fs-CBD), compared to Broad-Spectrum CBD (bs-CBD) and placebo, reduce participant alcohol consumption?
* Does Full-Spectrum CBD (fs-CBD), compared to Broad-Spectrum CBD (bs-CBD) and placebo, reduce negative emotionality and other AUD phenotypes?
* What are the effects of fs-CBD and bs-CBD on the gut microbiome and gut permeability?

Researchers will compare fs-CBD to bs-CBD and a placebo (a look-alike substance that contains no CBD or THC) to see if fs-CBD reduces participant alcohol consumption.

Participation will last 12 weeks during which participants will:

* Take the randomly assigned study drug (fs-CBD, bs-CBD, or placebo) daily for 8 weeks and report alcohol use via daily surveys
* Attend 5 in-person study visits
* Check in virtually with study staff weekly during the 8-week medication period

DETAILED DESCRIPTION:
This project is a randomized, placebo-controlled trial comparing the effects of Full-Spectrum CBD ([fs-CBD] CBD with < .03% THC) relative to Broad-Spectrum CBD ([bs-CBD] CBD that does not contain THC) and placebo, on alcohol consumption (in the lab and in the real world [Aim 1]) and on several clinically relevant Alcohol Use Disorder (AUD) phenotypes (Aims 2 and 3), among adults with AUD. Specifically, this trial will test the effects of fs-CBD (vs. bs-CBD and placebo) on self-reported alcohol intake over a 12-week period, alcohol self-administered during a session in our bar lab, and an alcohol biomarker in the blood over the course of the 12-week study. Investigators will also test the effects of fs-CBD (vs. bs-CBD and placebo) on a battery of AUD phenotyping measures (corresponding to the Addictions Neuroclinical Assessment [ANA] domains) that could aid in identifying individuals for whom fs-CBD is likely to be an effective treatment (Aim 2) and on the gut microbiome (Exploratory Aim 3), which has been shown to play an important role in the etiology and maintenance of AUD. Investigators will recruit adults with AUD to be randomly assigned to take 200 mg of fs-CBD, bs-CBD, or placebo daily for 8 weeks. During this 8-week period, participants will report alcohol use via daily surveys and have weekly, virtual check-ins with study staff. Subjects will attend five in-person study sessions, provide two home-collected fecal samples for assaying the gut microbiome, and have blood drawn several times to measure CBC, CMP, PEth, gut permeability, and blood cannabinoid levels throughout the study. At the end of the 8-week study medication period, participants will attend a lab session involving an alcohol self-administration (bar lab) task, ANA assessments, and a blood draw (to measure an alcohol biomarker and circulating gut markers). The ANA battery and blood and fecal samples will also be collected prior to starting study medication, so that post-intervention change in the proposed mediators can be measured. Study participation will span 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 21-65
2. Provides informed consent to participate
3. Meets the following cannabis use criteria:

   * Are not CBD or THC naïve: have used CBD or a cannabis product containing CBD at least once in the last year and have used THC or a cannabis product containing THC at least once in the last year
   * Are not frequent cannabis users (those who use cannabis 6 or more times per month over the past 3 months will be excluded)
4. Meets Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) criteria for current Alcohol Use Disorder (AUD) of at least moderate severity (i.e., 4 or more DSM-V symptoms)
5. Meets the following drinking criteria:

   * Must have consumed alcohol at least 2x per week, with a minimum of 20 drinks per week (for both males and females), consistently for the past three months.
   * Must report at least 1 heavy drinking day per week over the past 3 months (5 or more drinks per day for males, 4 or more drinks per day for females)
6. Willing to provide fecal samples
7. Willing to have their blood drawn
8. Able to attend in-person visits at the study site

Exclusion Criteria:

1. Must not currently take any of the following medications:

   * Those known to have a major interaction with Epidiolex
   * Those known to have a major interaction with Marinol
   * Acute treatment with any antiepileptic medications
   * Acute treatment with any psychotropic medications besides antidepressants (Note participants using antidepressants must be on a stable dose for the past 90 days and should not require medication adjustments during the study period. Those who do not meet these criteria will be excluded).
   * Medication known to affect alcohol intake (e.g., disulfiram, naltrexone, acamprosate, and/or topiramate, etc.)
2. Females must not be pregnant, nursing, nor planning a pregnancy. Individuals not using contraception or practicing abstinence will also be excluded
3. Must not be positive for any illicit drugs (besides cannabis) on urine drug screen or self- report any illicit/recreational drug use in the past 30 days.
4. Must not have a history of a serious DSM-V psychiatric disorder, including bipolar affective disorder, schizophrenia, cluster B personality disorders (borderline, antisocial, histrionic, narcissistic), or any other psychotic mental disorder. Must not have a current diagnosis of an eating disorder, panic disorder, obsessive/compulsive disorder, or post-traumatic stress disorder.
5. Must not meet criteria for a medical condition that contraindicates the use of CBD
6. Must not have clinically significant medical problems in the last six months, such as cardiovascular, renal, gastrointestinal, or endocrine problems, that would impair participation or limit medication ingestion
7. Must not report a history of alcohol-related liver disease or alcohol-related medical illness, such as gastrointestinal bleeding, pancreatitis, hepatocellular disease, or peptic ulcer

   • We will evaluate hepatocellular disease throughout the study (Baseline, Week 4, Week 8, and Week 12 Visits), subjects with elevations of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than two times the upper limit of the normal range will be withdrawn and referred for medical treatment.
8. Must not have used antibiotics in the past three months
9. Must not have ever been diagnosed with a gastrointestinal disorder
10. Must not have used probiotic supplements in the past one month.
11. Must not be seeking treatment/in treatment for AUD or another substance use disorder.
12. Must not have a history of severe alcohol withdrawal (e.g., seizure, delirium tremens)

    • Assessed via self-report during screening and with the Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) at the Baseline, Medication Dispense, Week 4, Week 8, and Week 12 study visits. Subjects who score greater than 7 on the CIWA-Ar will be withdrawn and referred for medical treatment.
13. Must not have a current diagnosis of a substance use disorder besides AUD (note: cannabis use disorder is also exclusionary)
14. Current suicidality risk as indicated during the conduct of the C-SSRS with concurrence after a study physician's or PI evaluation if the response to C-SSRS questions 1 or 2 is "yes"

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol Self-Administration During the Bar Lab Task | Week 8
  Number of drinks (between 0-8) subjects choose to self-administer during the Bar Lab Alcohol Self-Administration Task at the week 8 study visit.
Change in Self-Report of Drinking Behavior (Drinks Per Drinking Day) | Baseline, Week 4, Week 8, and Week 12
  Drinks Per Drinking Day (DPDD) during the 12-week study period as reported on Timeline Follow Back at Baseline (prior to treatment), Week 4, Week 8, and Week 12.
Change in Phosphatidylethanol (PEth) | Baseline, Week 4, Week 8, and Week 12
  Phosphatidylethanol (PEth) concentration in blood samples collected at Baseline (prior to treatment), Week 4, Week 8, and Week 12.

SECONDARY OUTCOMES:
Change in Negative Emotionality ANA Domain Score | Baseline, Week 8
  This summary score will be calculated for change from baseline to follow-up for each of the four ANA Negative Emotionality Measures (Beck Depression Inventory-II, Beck Anxiety Inventory, State-Trait Anxiety Inventory and Drinker Inventory of Consequences-2R) . We will first subtract baseline raw scores from follow-up raw scores for each measure. The summary score will be comprised of the average of the standardized Z scores of the change scores created for each of the four measures. Z scores will range from -3 to 3 after adjusting for outliers, with higher average Z scores indicating a worse outcome.

OTHER OUTCOMES:
Change in Gut Microbial Diversity | Baseline, Week 8
  Gut microbial diversity from fecal samples collected at Baseline (prior to treatment) and Week 8.
Change in Gut Permeability (Lipopolysaccharide Binding Protein [LBP]) | Baseline, 8 Weeks
  Lipopolysaccharide Binding Protein levels in blood samples collected at Baseline (prior to treatment) and Week 8.
Change in Gut Permeability (CD14) | Baseline, 8 Weeks
  CD14 levels in blood samples collected at Baseline (prior to treatment) and Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Hollis C Karoly, PhD, Principal Investigator — University of Colorado School of Medicine- Anschutz Medical Campus
Locations (1):
- University of Colorado School of Medicine- Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will submit all de-identified individual level phenotypic human subjects data from this project to the National Institute on Alcohol Abuse and Alcoholism (NIAAA) Data Archive, which is part of the National Institutes of Mental Health (NIMH) Data Archive (NDA).
  The project also involves collection of human specimens (fecal samples) which will generate non-human genomic data. Specifically, investigators plan to generate 360 (180 subjects x 2 timepoints) human gut microbiota metagenomes (i.e., gut microbiome). Deidentified genomic data (microbiome sequencing from the fecal samples) will be uploaded to the appropriate data repository upon NIH program administrator determination (NDA or the database of Genotypes and Phenotypes [dbGaP]).
  Participants will be given the option in the consent/HIPAA form to allow the use of any leftover samples to bank for future undetermined analyses not specified in the protocol.
Supporting Information: Study Protocol, SAP
Time Frame: Human phenotypic data will be uploaded at least twice a year, following NIMH Data Archive (NDA) requirements. Non-human genomes from fecal samples will be shared within 12 months of processing and genotyping all meta-genomes.
Access Criteria: Data access will be through the National Institute of Mental Health Data Archive (NDA) and/or the database of Genotypes and Phenotypes (dbGaP).